CLINICAL TRIAL: NCT04777565
Title: The Efficacy of a Minimally Invasive Direct Cochlear Access Via the HEARO Procedure
Brief Title: Study of a Minimally Invasive Cochlear Access for Cochlear Implantation Via a Robotic Procedure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: MED-EL Elektromedizinische Geräte GesmbH (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: MED-EL_HEARO_french_study
Record Dates: First submitted 2021-02-10; First posted 2021-03-02 (Actual); Last update posted 2023-02-21 (Actual); Status verified 2023-02

CONDITIONS: Sensorineural Hearing Loss, Bilateral
Keywords: cochlear implant; robotic surgery; electrode insertion
MeSH Terms: conditions — Hearing Loss, Sensorineural | interventions — Robotic Surgical Procedures

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CI surgery (Experimental): cochlear implant surgery
  Interventions: Other: Robotic surgery

INTERVENTIONS:
Other: Robotic surgery — Cochlear implant surgery with HEARO procedure

SUMMARY:
The objectives of this study are to explore the efficacy and safety of a robotic procedure for a minimally invasive cochlear implantation.

DETAILED DESCRIPTION:
The cochlear implant (CI) is a neural prothesis and has been the gold standard treatment for severe to profound sensorineural hearing loss over several decades. The surgical procedure for cochlear implantation surgery aims to atraumatically insert the electrode array of the cochlear implant into the cochlea. However, due to the location of the cochlea inside the skull, the surgeon is required to initially create an access from the surface of the temporal bone to the cochlea (inner ear). In conventional methods, this access is acquired by removal of large portions of the mastoid bone through a wide mastoidectomy and posterior tympanotomy. The outcome and success of the conventional procedure varies due to mainly two factors: surgeon skill and subject anatomical variation.

To overcome these variables toward a more consistent and less invasive cochlear implantation surgery, the development of robotic and image guided cochlear implantation has taken place.

This study primarily aims to explore the efficacy of the HEARO robotic cochlear implantation surgery.

Primary Objective

The primary objective of this study is to:

• explore the efficacy of a minimally invasive direct cochlear access via the HEARO procedure.

Secondary Objectives

The secondary objectives of this study are to:

* explore the safety of a minimally invasive direct cochlear access via the HEARO procedure.
* exploratively evaluate the electrode array insertion outcomes through the direct tunnel access.

ELIGIBILITY:
Inclusion Criteria:

* Subjects scheduled for CI surgery according to clinical routine
* Subjects who will receive a cochlear implant of the MED-EL portfolio
* Signed and dated informed consent form

Exclusion Criteria:

* Lack of compliance with any inclusion criteria
* Age under 18 years
* Pregnancy
* Distance of the planned trajectory to the facial nerve is < 0.4 mm as per screening CT scan
* Distance of the planned trajectory to the chorda tympani is < 0.3 mm as per screening CT scan
* A safe inner ear access cannot be planned for preservation of RW membrane and cochlear structures
* Individuals where image guidance or robotic procedures are not indicated
* Individuals who have known allergy to components of the cochlear implant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2021-09-15 (Actual); Primary Completion 2023-01-01 (Actual); Study Completion 2023-01-01 (Actual)

PRIMARY OUTCOMES:
Electrode array insertion | During surgery
  • Relative ratio of successful electrode array insertions through the drilled direct cochlear access with the HEARO procedure to the total HEARO procedures (i.e. proportion of successful insertions with the procedure out of the total number of patients included in the study).

SECONDARY OUTCOMES:
Electrode array insertion outcome (efficacy) | During surgery
  • The angular insertion depth will be evaluated.
Electrode array insertion outcome (efficacy) | During surgery
  • The number of contacts inserted will be evaluated.
Electrode array insertion outcome (efficacy) | During surgery
  • The tip-fold over will be evaluated.
Electrode array insertion outcome (efficacy) | During surgery
  • The scalar deviation will be evaluated.
Insertion depth prediction accuracy (efficacy) | During surgery
  • The insertion depth prediction accuracy as the difference between the estimated insertion depth of the electrode at the planning and the actual insertion depth.
Absolute angular accuracy of the drilled tunnel access (safety) | During surgery
  • The absolute lateral accuracy of the drilled tunnel to the facial nerve and chorda tympani is measured as the difference between the planned trajectory and the actual drilled trajectory distance.
Absolute lateral accuracy of the drilled tunnel at the target (safety) | During surgery
  • The absolute lateral accuracy of the drilled tunnel is measured as the distance between the planned target trajectory position and actual target of the drilled trajectory position.
Ratio of the round window membrane preservation during the inner ear access (safety) | During surgery
  • The ratio of the preserved round window (RW) membrane at the robotic inner ear access by visual inspection. This will be assessed as subjective evaluation by the surgeon.
Timing of the HEARO procedure | During surgery
  • The timing of the different steps of the HEARO procedure will be recorded.
Adverse events (safety) | During surgery
  • Adverse events will be recorded

CONTACTS AND LOCATIONS:
Overall Officials: Frédéric Venail, Pr, Principal Investigator — University Hospital, Montpellier
Locations (1):
- CHU Montpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Fourez AL, Kaderbay A, Villerabel C, Korchagina J, Pean V, Mondain M, Venail F. Implementation of Robot-Assisted Minimally Invasive Cochlear Implantation: A Feasibility Study. Otol Neurotol. 2025 Aug 1;46(7):809-815. doi: 10.1097/MAO.0000000000004531. Epub 2025 May 23. PMID 40423721